CLINICAL TRIAL: NCT06462872
Title: To Study the Efficacy of Intravenous Neostigmine in Resolution of Acute GI Paralysis in Critically Ill Cirrhotics-Prospective Observational Study
Brief Title: To Study the Efficacy of Intravenous Neostigmine in Resolution of Acute GI Paralysis in Critically Ill Cirrhotics
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-66
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Critically Ill Cirrhotics
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill cirrhotics: Critically ill cirrhosis patient admitted in liver ICU with new onset acute GI tract paralysis and develop feed intolerance.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — It is an observational study

SUMMARY:
Aim: To determine the efficacy of intravenous neostigmine in the resolution of acute GI paralysis in patients with Critically Ill Cirrhosis (CIC).

Study population: Critically ill cirrhosis patient admitted in liver ICU with new onset acute GI tract paralysis and develop feed intolerance.

Study period - 1 years Sample Size

• All the consecutive patients admitted in liver ICU during the study time period (Dec 2023 -September 2024) will be screened and those patients meeting with inclusion and exclusion criteria will be enrolled, we intend to enroll 70 patients for the study.

DETAILED DESCRIPTION:
Study Design: Prospective observational study

Intervention: Standard medical treatment (SMT)- keeping patients Nil Per Oral, I.V fluids, I.V antibiotics (antibiotic as per ICU protocol of ILBS), Ryle's tube decompression, correction of dyselectrolytemia, prokinetics

* Patient to receive slow intravenous infusion of Neostigmine, 1 mg over 5-10 minutes repeated 8 hourly for first 24 hours.
* Administration of Neostigmine will include defined steps for prevention of adverse event:

  * Neostigmine, 1 mg, intravenous infusion over 3-5 min
  * Atropine available at bedside Patient kept supine
  * Continuous electrocardiographic monitoring with vital signs for30 min
  * Continuous clinical assessment for 15-30 min

Patients who do not give consent for the intervention will receive the standard of care treatment.

Rescue treatment- Colonoscopic decompression, Flatus tube insertion, surgical intervention

Monitoring and assessment:

. An immediate clinical response was defined as the passage of flatus or stool with reduction in abdominal distention on physical examination after the injection. With clinical and radiological confirmation of resolution and re-initiation of enteral feeding, would define clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill cirrhosis patient admitted in liver ICU with new onset acute GI tract paralysis and develop feed intolerance.
2. Patients with new onset lower GI tract paralysis with clinical presentation of feed intolerance defined as GRV> 500ml, abdominal distension, bowel distension on abdominal imaging, and absence of bowel sounds.

Exclusion Criteria:

1. Recent GI bleed
2. Bronchoconstriction
3. Bradycardia
4. Current or past history of surgical abdomen, including mechanical obstruction, mesenteric ischemia, perforation or requiring abdominal surgery.
5. Prior comorbid illnesses like advanced cardiopulmonary disease, prior episodes of arrhythmia, structural heart diseases, traumatic brain injury, cerebrovascular accidents, raised intracranial pressures, history of myasthenia gravis.
6. Endocrinological illnesses like uncontrolled hypothyroidism, hypoparathyroidism
7. Connective tissue disorders including systemic sclerosis, dermatomyositis or polymyositis, systemic lupus erythematosus,amyloidosis.
8. Pregnant females
9. Refusal to give consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill cirrhosis patient admitted in liver ICU with new onset acute GI tract paralysis and develop feed intolerance.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
To study the proportion of patients reinitiated on enteral nutrition within 24 hours after radiological resolution. | 24 hours

SECONDARY OUTCOMES:
Proportion of patients having passage of stool after intravenous neostigmine within 24-hours. | 24 hours
Time to passage of stool in between two groups. | 7 days
Change in intra-abdominal pressure after resolution (IAP before and after) | 7 days
Serial change in gastric residual volumes (GRV) | 7 days
Calorie intake in 7 days | 7 days
Change in SOFA score. | 7 days
Change in APACHE score | 7 days
Number of patients with new onset organ failure | 7 days
Number of patients with new onset SBP | 7 days
Number of patients with new onset infections | 7 days
Number of patients with need for rescue treatment. | 7 days
Proportion of patients showing radiological resolution within 48-Hours and 72- hours. | within 48-Hours and 72- hours
Adverse effects related to the treatment and need for atropine usage. | 7 days
Survival at 7-days | 7 days
Stool microbiome study based on 16S RNA sequencing (Sample willbe stored in bio-bank). | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided